CLINICAL TRIAL: NCT02254187
Title: A Randomised, Open-label Three-way Crossover Study to Evaluate the Pharmacokinetics of Salmeterol After Inhalation of a 25 μg and 50 μg Single Dose (Inhalation Powder, Hard PE Capsule for HandiHaler®2) and a 50 μg Single Dose (Serevent® Diskus®) in Healthy Male Volunteers
Brief Title: Pharmacokinetics of Salmeterol Via HandiHaler® in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1184.17
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — Salmeterol Xinafoate

ARMS (3):
- Salmeterol capsule via Handihaler - low (Experimental)
  Interventions: Drug: Salmeterol capsule - low
- Salmeterol capsule via Handihaler - high (Experimental)
  Interventions: Drug: Salmeterol capsule - high
- Salmeterol via Serevent® Diskus® (Active Comparator)
  Interventions: Drug: Salmeterol via Serevent® Diskus®

INTERVENTIONS:
Drug: Salmeterol capsule - low
  Arms: Salmeterol capsule via Handihaler - low
Drug: Salmeterol capsule - high
  Arms: Salmeterol capsule via Handihaler - high
Drug: Salmeterol via Serevent® Diskus®
  Arms: Salmeterol via Serevent® Diskus®

SUMMARY:
The objective of this study is to investigate if the systemic drug exposure of at least 25 μg and perhaps 50 μg salmeterol presented as inhalation powder in PE capsules and administered via HandiHaler® 2 does not exceed that of 50 μg Serevent® Diskus® and to investigate safety and tolerability of salmeterol presented as inhalation powder in PE capsules and administered via HandiHaler® 2

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male based upon a complete medical history, including the physical examination, regarding vital signs ((Blood Pressure (BP), Pulse Rate (PR)), 12-lead ECG measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease.
2. Age ≥21 and ≤50 years
3. BMI ≥18.5 and <30 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

1. Any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
2. Evidence of a clinically relevant concomitant disease
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
4. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to randomization
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to randomization
10. Participation in another trial with an investigational drug within 2 months prior to randomization
11. Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
12. Inability to refrain from smoking on trial days as judged by the investigator
13. Alcohol abuse (more than 60 g alcohol a day)
14. Drug abuse
15. Blood donation (more than 100 mL blood within 4 weeks prior to randomization or during the trial)
16. Excessive physical activities within 1 week prior to randomization or during the trial
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of the study centre

    The following exclusion criteria are specific for this study due to the known class side effect profile of ß2-mimetics:
19. Asthma or history of pulmonary hyperreactivity
20. Hyperthyrosis
21. Allergic rhinitis in need of treatment
22. Clinically relevant cardiac arrhythmia
23. Paroxysmal tachycardia (>100 beats per minute)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of salmeterol in blood plasma over the time interval from 0 extrapolated to infinity) | up to 8 hours after drug administration
Cmax (maximum measured concentration of salmeterol in blood plasma) | up to 8 hours after drug administration

SECONDARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of salmeterol in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 8 hours after drug administration
AUCt1-t2 (area under the concentration time curve of salmeterol in plasma over the time interval t1 to t2) | up to 8 hours after drug administration
tmax (time from dosing to the maximum concentration of salmeterol in plasma) | up to 8 hours after drug administration
λz (terminal rate constant in plasma) | up to 8 hours after drug administration
t½ (terminal half-life of salmeterol in plasma) | up to 8 hours after drug administration
MRTih (mean residence time of salmeterol in the body after inhalational administration) | up to 8 hours after drug administration
CL/F (apparent clearance of salmeterol in the plasma after extravascular administration) | up to 8 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase (λz) following an extravascular dose) | up to 8 hours after drug administration
Number of patients with abnormal changes in laboratory parameters | up to 14 days following the last drug administration
Number of patients with clinically significant changes in vital signs | up to 14 days following the last drug administration
  Blood Pressure, Pulse Rate
Number of patients with clinically significant changes in 12-lead ECG parameters | up to 14 days following the last drug administration
Number of patients with adverse events | up to 14 days following the last drug administration
Assessment of tolerability by investigator on a 4-point scale | 14 days following the last drug administration